CLINICAL TRIAL: NCT04034017
Title: Personal, Academic and Stress Correlates of Gastroesophageal Reflux Disease Among College Students in Southwestern Saudi Arabia: A Cross-sectional Study
Brief Title: Gastroesophageal Reflux Disease Among College Students
Status: Completed | Type: Observational
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Nabil Awadalla, Principal investigator, King Khalid University
Other Study IDs: ECM
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Gastroesophageal Reflux
Keywords: College students; Gastroesophageal reflux disease; GERD; Prevalence; Perceived stress
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — descriptive study, no intervention

SUMMARY:
Background: Gastroesophageal reflux disease (GERD) is a worldwide prevalent gastrointestinal disorder which has negative impacts on quality of life, health and economy. The aims of this study were to assess the prevalence of GERD among college students in southwestern Saudi Arabia and to evaluate its personal, academic and stress correlates Materials and Methods: Through a cross-sectional study design, a self-reported questionnaire was distributed between a representative sample of students in health and non-health care colleges in southwestern Saudi Arabia. The questionnaire included data for personal characteristics, academic study, and Arabic versions of GERD questionnaire (GerdQ) and Cohen's Perceived Stress Scale.

DETAILED DESCRIPTION:
Study design and setting A cross-sectional study was carried out in both male and female campuses of King Khalid University (KKU) during the academic year 2018-2019. The University is located in Aseer region in the southwestern part of Saudi Arabia. The area of Aseer region is about 80.000 square kilometers occupied with more than 1.6 million people. The university comprise 5 health colleges and 24 non-health colleges with a total number of 60.312 male and female students in the academic year 2014-2015.

Target population Students in Health and non-health care colleges in KKU were the target population.

Sample size and sampling method Sample size was estimated by using Epi info program version 7.2 with the anticipated prevalence of GERD symptoms among college students 23.8% [6], 95% confidence level and acceptable margin of error of 2.5%. The calculated cluster size was 1113 students. To account for the possibility of non-response, 1200 students were targeted from each of health and non-health care colleges.

All health care colleges were included in the study. They were colleges of medicine, pharmacy, dentistry, nursing and applied medical science. Five non- health care colleges were selected by random method. They were colleges of education, science, humanities, administrative and financial sciences, and languages and translation. Participants were selected through stratified cluster sampling technique. Within each college, students were stratified by academic level. Within each level a cluster (section or study group) was selected. When possible, all registered students within each cluster were included.

Study tool and data collection A self-reported questionnaire was distributed personally by medical students-during their training in community medicine course- between the participants. The questionnaire includes the following sections: a) personal data such as, age sex, marital status, smoking status and family income; b) academic data which include, name of college, academic level and Grade point average (GPA); c) Arabic version of GERD questionnaire (GerdQ)[10]; d) Arabic version of Cohen's Perceived Stress Scale (PSS) [8].

All incomplete questionnaires were excluded. Arabic version of GERD questionnaire (GerdQ) GerdQ is a valid questionnaire used to explore the probaility of GERD. It is consisted of 6 questions as follow: four positive questions to assess GERD symptoms (heartburn, regurgitation, sleep disturbance related to heartburn and regurgitation and use of medications) and two negative questions (epigastric pain and nausea). Each item rated from 0 to 3 depending on the rate of symptoms over the previous week. GERD was detected with a total score value of 8 or more [10]. Score value of 8 or more plus total score value of 3 or more for the impact questions (sleep disturbance and use of medications) indicted GERD with impact on daily life. The Arabic version of GerdQ was developed and validated for use among Arabic speakers [11].

Data analysis The gained data were entered, revised, and analyzed using SPSS, version 22 software package. Grading of PSS into low, moderate and high was according to Cohen's et al [12]. Crude odds ratio (cOR) and adjusted odds ratio (aOR) were calculated using univariate and multivariable logistic regression analysis respectively. Their 95% confidence intervals (95% CIs) were used to identify significant factors associated with GERD among students.

ELIGIBILITY:
Inclusion Criteria:

* College students
* Must be cooperative
* Agree to participate

Exclusion Criteria:

* non cooperative students
* disagree to participate in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A representative sample of Students in Health and non-health care colleges in King Khalid U
Sampling Method: Probability Sample
Enrollment: 2878 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
prevalence rate of gastroesophogeal reflux disease (GERD) among college students | 1 year
  Arabic version of GERD questionnaire (GerdQ) was used to screen for GERD among college students. GERD was considered with a total score value of GerdQ of 8 or more
assess the association of GERD with students' personal data | 1 year
  examining the associations of GERD with the personal data such as, age (in years) sex (male Vs. female), marital status (married Vs. single), smoking status (smoker, ex-smoker and non-smoker) and family income (sufficient Vs. insufficient)
assess the association of GERD with students' academic data | 1 year
  the academic data include: college(health care Vs. non-health care colleges) academic year (first year through six year) student's Grade point average (GPA) in the previous academic year
examine the association of GERD with the level of perceived stress | 1 year
  perceived stress was assessed by using the Arabic version of Cohen's Perceived Stress Scale (PSS). Grading of PSS into low, moderate and high was done as the following: scores ranging from 0-13 was considered low stress; scores ranging from 14-26 was considered moderate stress; scores ranging from 27-40 was considered high perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid University, Abhā, 'Asir Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No